CLINICAL TRIAL: NCT01607411
Title: A Clinical Study to Evaluate Experimental Children's Toothpastes in an In-Situ Caries Model
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RH01390
Record Dates: First submitted 2012-02-16; First posted 2012-05-30 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Fluorides

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fluoride free toothpaste (Placebo Comparator): toothpaste with no fluoride
  Interventions: Drug: Placebo
- 1426ppm Fluoride Toothpaste (Experimental): Experimental toothpaste containing 1426 ppm Fluoride
  Interventions: Drug: Fluoride
- 1000 ppm Fluoride Toothpaste (Experimental): Experimental toothpaste containing 1000 ppm Fluoride
  Interventions: Drug: Fluoride
- 500 ppm Toothpaste (Experimental): Experimental toothpaste containing 500 ppm Fluoride
  Interventions: Drug: Fluoride

INTERVENTIONS:
Drug: Fluoride — Fluoride Toothpaste
  Arms: 1000 ppm Fluoride Toothpaste; 1426ppm Fluoride Toothpaste; 500 ppm Toothpaste
Drug: Placebo — Fluoride free toothpaste
  Arms: Fluoride free toothpaste

SUMMARY:
An in situ model will be used to evaluate and compare enamel remineralization of human enamel specimens after single use of experimental children's toothpastes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 11 to 14 inclusive who have an unstimulated salivary flow rate of at least 0.2 mL/minute and a stimulated salivary flow rate of at least 0.8 mL/minute (Screening Visit 1).

Exclusion Criteria:

-

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Newby EE, Martinez-Mier EA, Hara A, Lippert F, Kelly SA, Fleming N, Butler A, Bosma ML, Zero DT. A randomised clinical study to evaluate experimental children's toothpastes in an in-situ palatal caries model in children aged 11-14 years. Int Dent J. 2013 Dec;63 Suppl 2(Suppl 2):31-8. doi: 10.1111/idj.12073. PMID 24283282

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of the 70 participants screened, 15 were not randomized into the study (12 did not meet study criteria and 3 withdrew the consent). A washout fluoride (F) toothpaste was used for a week prior treatment. In-situ appliances were prepared for participants to fit enamel specimens.
Groups:
- Sodium Fluoride(NaF) Toothpaste (1426parts Per Million(Ppm) F): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.0 grams (g) ± 0.1g of NaF toothpaste(1426 ppm F) and expectorated. The direct contact between palatal appliance and toothbrush was avoided
- NaF Toothpaste (1000 Ppm F): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.0 g ± 0.1g of NaF toothpaste (1000 ppm F) and expectorated. The direct contact between palatal appliance and toothbrush was avoided
- NaF Toothpaste (500 Ppm F): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.0 g ± 0.1g of NaF toothpaste (500 ppm F) and expectorated. The direct contact between palatal appliance and toothbrush was avoided
- Placebo Toothpaste (0 Ppm F): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.0 g ± 0.1g of NaF toothpaste (0ppm F) and expectorated. The direct contact between palatal appliance and toothbrush was avoided
Period: Period I
Arm/Group | Sodium Fluoride(NaF) Toothpaste (1426parts Per Million(Ppm) F) | NaF Toothpaste (1000 Ppm F) | NaF Toothpaste (500 Ppm F) | Placebo Toothpaste (0 Ppm F)
Started | 14 | 13 | 14 | 14
Completed | 14 | 13 | 14 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Period II
Arm/Group | Sodium Fluoride(NaF) Toothpaste (1426parts Per Million(Ppm) F) | NaF Toothpaste (1000 Ppm F) | NaF Toothpaste (500 Ppm F) | Placebo Toothpaste (0 Ppm F)
Started | 14 (Due to crossover design, different set of participants entered Period 2) | 14 (Due to crossover design, different set of participants entered Period 2) | 13 (Due to crossover design, different set of participants entered Period 2) | 14 (Due to crossover design, different set of participants entered Period 2)
Completed | 14 | 14 | 13 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Period III
Arm/Group | Sodium Fluoride(NaF) Toothpaste (1426parts Per Million(Ppm) F) | NaF Toothpaste (1000 Ppm F) | NaF Toothpaste (500 Ppm F) | Placebo Toothpaste (0 Ppm F)
Started | 14 (Due to crossover design, different set of participants entered Period 3) | 14 (Due to crossover design, different set of participants entered Period 3) | 14 (Due to crossover design, different set of participants entered Period 3) | 13 (Due to crossover design, different set of participants entered Period 3)
Completed | 14 | 14 | 14 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Period IV
Arm/Group | Sodium Fluoride(NaF) Toothpaste (1426parts Per Million(Ppm) F) | NaF Toothpaste (1000 Ppm F) | NaF Toothpaste (500 Ppm F) | Placebo Toothpaste (0 Ppm F)
Started | 13 (Due to crossover design, different set of participants entered Period 4) | 14 (Due to crossover design, different set of participants entered Period 4) | 14 (Due to crossover design, different set of participants entered Period 4) | 14 (Due to crossover design, different set of participants entered Period 4)
Completed | 13 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All randomized participants who received atleast one dose of the study treatments
Arm/Group | Overall
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.4 (1.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 9
  White | 41
  More than one race | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage Surface Microhardness Recovery of Test Dentifrices Relative to Placebo Dentifrice
Description: Surface microhardness recovery (SMHR) test was used to assess the changes in mineralization status of enamel specimens using a Wilson 2100 Hardness tester. SMHR was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents rehardening of enamel surface. Percent SMHR was calculated from indentation values of enamel specimens at baseline (B), after in-situ hardening (R) and after first demineralization challenge (D1) using formula: [(D1-R)/ (D1-B)]*100.
Time Frame: Baseline to 4 hours
Population: Per Protocol (PP) Population: All randomized participants who received at least one study product, had one efficacy assessment and did not have any protocol violations deemed to affect efficacy. Missing enamel specimen values were imputed, by averaging over the available enamel specimens.
Measure: Mean (Standard Error); unit: %SMHR
Groups:
- NaF Toothpaste (1426 Ppm F): Participants were fitted with enamel specimen appliance in the palatal surface 5 minutes before treatment initiation. Participants brushed their teeth for one timed minute with 1.0 g ± 0.1g of NaF toothpaste (1426 ppm F) and expectorated. The direct contact between palatal appliance and toothbrush was avoided
Arm/Group | NaF Toothpaste (1426 Ppm F) | NaF Toothpaste (1000 Ppm F) | NaF Toothpaste (500 Ppm F) | Placebo Toothpaste (0 Ppm F)
Number analyzed (Participants) | 55 | 55 | 55 | 55
%SMHR | 30.72 (0.87) | 29.49 (0.87) | 28.29 (0.87) | 25.13 (0.87)
Statistical Analysis 1: Comparison: NaF Toothpaste (1426 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 5.59, 95% CI 2-sided [3.60 to 7.58] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: NaF Toothpaste (1000 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 4.36, 95% CI 2-sided [2.37 to 6.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF Toothpaste (500 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p = 0.0021, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 3.16, 95% CI 2-sided [1.17 to 5.15] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: %SMHR of Enamel Specimens Exposed to Test Treatments
Description: as for outcome 1
Time Frame: Baseline to 4 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: %SMHR
Arm/Group | NaF Toothpaste (1426 Ppm F) | NaF Toothpaste (1000 Ppm F) | NaF Toothpaste (500 Ppm F)
Number analyzed (Participants) | 55 | 55 | 55
%SMHR | 30.72 (0.87) | 29.49 (0.87) | 28.29 (0.87)
Statistical Analysis 1: Comparison: NaF Toothpaste (1426 Ppm F) vs NaF Toothpaste (1000 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p = 0.2225, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 1.23, 95% CI 2-sided [-0.76 to 3.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF Toothpaste (1426 Ppm F) vs NaF Toothpaste (500 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p = 0.0168, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 2.44, 95% CI 2-sided [0.44 to 4.43] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF Toothpaste (1000 Ppm F) vs NaF Toothpaste (500 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p = 0.2352, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 1.20, 95% CI 2-sided [-0.79 to 3.19] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percent Net Acid Resistance (%NAR) of Enamel Specimens
Description: Changes in mineral content of enamel specimens exposed to dietary erosive challenge were determined by measuring the length of the indentations. Decrease in the indentation length compared to the baseline indicates hardening of enamel surface. Enamel specimens were exposed to second erosion challenge to determine NAR which compared the indentations values of sound enamel specimens at baseline (B), first demineralization challenge (D1) and second demineralization challenge (D2). Percent NAR was calculated by formula: [(D1-D2)/ (D1-B)]*100.
Time Frame: Baseline to 4 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: %NAR
Arm/Group | NaF Toothpaste (1426 Ppm F) | NaF Toothpaste (1000 Ppm F) | NaF Toothpaste (500 Ppm F) | Placebo Toothpaste (0 Ppm F)
Number analyzed (Participants) | 55 | 55 | 55 | 55
%NAR | -19.72 (1.90) | -19.52 (1.90) | -25.82 (1.90) | -54.38 (1.90)
Statistical Analysis 1: Comparison: NaF Toothpaste (1426 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 34.65, 95% CI 2-sided [30.07 to 39.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF Toothpaste (1000 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean difference = 34.86, 95% CI 2-sided [30.28 to 39.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF Toothpaste (500 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 28.55, 95% CI 2-sided [23.97 to 33.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: NaF Toothpaste (1426 Ppm F) vs NaF Toothpaste (1000 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p = 0.9292, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = -0.21, 95% CI 2-sided [-4.79 to 4.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: NaF Toothpaste (1426 Ppm F) vs NaF Toothpaste (500 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p = 0.0094, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 6.10, 95% CI 2-sided [1.52 to 10.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: NaF Toothpaste (1000 Ppm F) vs NaF Toothpaste (500 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p = 0.0073, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 6.31, 95% CI 2-sided [1.72 to 10.89] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Enamel Fluoride Uptake
Description: Enamel fluoride uptake was determined using the microdrill enamel biopsy technique. The amount of fluoride uptake by enamel was calculated based on amount of F divided by volume of the enamel cores and expressed as micrograms (μg)* F/centimeters(cm)^2. Difference between treatments was calculated with respect to F uptake by enamel.
Time Frame: Baseline to 4 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: μg*F/cm^2
Arm/Group | NaF Toothpaste (1426 Ppm F) | NaF Toothpaste (1000 Ppm F) | NaF Toothpaste (500 Ppm F) | Placebo Toothpaste (0 Ppm F)
Number analyzed (Participants) | 55 | 55 | 55 | 55
μg*F/cm^2 | 1.76 (0.08) | 1.77 (0.08) | 1.47 (0.08) | 0.98 (0.08)
Statistical Analysis 1: Comparison: NaF Toothpaste (1426 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random factor; Adjusted Mean Difference = 0.78, 95% CI 2-sided [0.58 to 0.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF Toothpaste (1000 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 0.79, 95% CI 2-sided [0.58 to 0.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF Toothpaste (500 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 0.49, 95% CI 2-sided [0.29 to 0.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: NaF Toothpaste (1426 Ppm F) vs NaF Toothpaste (1000 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p = 0.9631, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = -0.005, 95% CI 2-sided [-0.21 to 0.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: NaF Toothpaste (1426 Ppm F) vs NaF Toothpaste (500 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p = 0.0047, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 0.29, 95% CI 2-sided [0.09 to 0.49] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: NaF Toothpaste (1000 Ppm F) vs NaF Toothpaste (500 Ppm F); Null hypothesis was no difference between treatments, being compared. Tests were 2 sided at 5% significance levels; Test type: Superiority or Other; p = 0.0040, ANOVA — No adjustment was required for multiple comparisons as the primary comparison was pre-specified; The fixed factors for ANOVA were study period and treatment and the subject was random effect; Adjusted Mean Difference = 0.30, 95% CI 2-sided [0.10 to 0.50] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline through 5 days post administration of last treatment
Arm/Group | NaF Toothpaste (1426 Ppm F) | NaF Toothpaste (1000 Ppm F) | NaF Toothpaste (500 Ppm F) | Placebo Toothpaste (0 Ppm F)
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 4/55 | 6/55 | 7/55 | 6/55
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaF Toothpaste (1426 Ppm F) (N=55) | NaF Toothpaste (1000 Ppm F) (N=55) | NaF Toothpaste (500 Ppm F) (N=55) | Placebo Toothpaste (0 Ppm F) (N=55)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Lip injury (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sinusitis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral herpes (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chapped lips (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival erythema (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.